CLINICAL TRIAL: NCT03457883
Title: Risk Factors for Recurrence After Pelvic Reconstruction of Pelvic Organ Prolapse：1 Year Follow-up in Patients Implanted Hernia Mesh and Biological Graft
Brief Title: Risk Factors for Recurrence After Pelvic Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xirong Guo, Vice President of Nanjing maternity and child Health Care Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NMU-2017323
Record Dates: First submitted 2018-02-26; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic organ prolapse; Vaginal mesh; biological graft; Recurrence
MeSH Terms: conditions — Pelvic Organ Prolapse; Recurrence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): accepted herniamesh mesh
  Interventions: Device: herniamesh
- group B (Experimental): accepted biological graft of cook
  Interventions: Device: biological graft

INTERVENTIONS:
Device: herniamesh — Patients were randomly assigned in a ratio of 1:1,by using SPSS19.0 statistical software, to either trocar-guided transvaginal mesh(herniamesh, group A) or biological graft (cook, group B)repair.
  Arms: group A
Device: biological graft — Patients were randomly assigned in a ratio of 1:1,by using SPSS19.0 statistical software, to either trocar-guided transvaginal mesh(herniamesh, group A) or biological graft (cook, group B)repair.
  Arms: group B

SUMMARY:
232 women underwent transvaginal mesh repair (TVM)with /without transvaginal hysterectomy for symptomatic POP, including group A（accepted herniamesh polypropylene mesh， 117 patients)；group B （underwent biological graft of cook，115 patients)；follow-ups for six months and one year after the surgery and a questionnaire about the life habits associated with relapse.

DETAILED DESCRIPTION:
We prospectively study a total of 232 women who underwent transvaginal mesh repair (TVM)with /without transvaginal hysterectomy for symptomatic POP, the patients into two groups :group A was accepted herniamesh polypropylene mesh(117)；group B underwent biological graft of cook(115)；Each patient underwent an interview that included a POP-Q which was quantified according to the Pelvic Organ Prolapse Quantitation (POPQ) system;follow-ups for six months and one year after the surgery and a questionnaire about the life habits associated with relapse.

ELIGIBILITY:
Inclusion Criteria:

242 postmenopausal patients with primary prolapse of the anterior vaginal wall or concomitant uterine prolapse,that was stage Ⅲ or higher (according to the Pelvic Organ Prolapse Quantification [POP-Q] system).

Exclusion Criteria:

pelvic floor repair surgery history and recurrent patients ; pelvic cancer and radiation to the pelvic area in the previous 6 months; simple uterine prolapse; combined with severe stress urinary incontinence or overactive bladder (OAB); local or systemic conditions that would preclude surgery or affect healing such as restricted leg motion (inability to conform to the lithotomy position) ; vaginal bleeding; infection; coagulation disorders; uncontrolled hypertension and diabetes mellitus;

Ages: 52 Years to 76 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
recurrence | at 12 months after surgery
  Recurrence was defined as a POP-quantification system stage ≥IIb or any symptomatic prolapse.

SECONDARY OUTCOMES:
perioperative complications | 12 months after surgery
  perioperative complications such as mesh exposure, extrusion , dyspareunia, urinary symptoms(New continence), pain (chronic pelvic pain and hip pain)